CLINICAL TRIAL: NCT02604758
Title: The Effect of the Psychiatric Nursing Approach Based on the Tidal Model on Coping and Self-esteem in People With Alcohol Dependency: A Randomized Trial
Brief Title: Tidal Model's Effect on Coping and Self-Esteem
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahire Olcay Çam (Other)
Responsible Party: Sponsor-Investigator, Mahire Olcay Çam, Faculty of Nursing, Ege University
Organization: Ege University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 7321
Record Dates: First submitted 2015-11-09; First posted 2015-11-13 (Estimated); Last update posted 2015-11-13 (Estimated); Status verified 2015-11

CONDITIONS: Alcoholism
Keywords: Alcoholics [M01.066]
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tidal Model (Experimental): the psychiatric nursing approach based on the Tidal Model
  Interventions: Behavioral: The Psychiatric Nursing Approach Based On The Tidal Model
- control group (No Intervention): The control group received routine treatment and follow-up in the Alcohol and Substance Addiction Treatment Clinic.

INTERVENTIONS:
Behavioral: The Psychiatric Nursing Approach Based On The Tidal Model — To provide individualized care for patients in the experimental group, the One-to-One Sessions were initiated and interventions were performed in line with the goals of the persons and the aims of the research. The interventions were selected from interventions regarding with coping and self-esteem from the Nursing Interventions Classification(NIC) system.The One-to-One sessions help the person recognize change and focus the person on achievement and goals.Taking into account the basic process of the Tidal Model, care stages, the following interview plan was drawn up, containing the details of the interviews to be carried out with people with alcohol dependency, and the One-to-One Sessions were held in line with this plan two times per week.
  Arms: Tidal Model

SUMMARY:
The aim of the study was to determine the effect of the psychiatric nursing approach based on the Tidal Model on coping and self-esteem in people with alcohol dependency.

ELIGIBILITY:
Inclusion Criteria:

* People with alcohol dependency were included in the study who were between 30 and 50 years of age who were admitted for treatment to the Alcohol and Substance Addiction Treatment clinic.

Exclusion Criteria:

* People with alcohol dependency who were severely depressed with a Beck Depression score of 41 or more and those with severe anxiety(a Beck Anxiety score of 26 or more) were not included in the study.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2013-10; Primary Completion 2014-09 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
The Coping Inventory | after three months
  The Coping Inventory was developed by Carver et al. in 1989, and Turkish validity and reliability were carried out in 2005 by Ağargün et al. Each sub-scale of COPE gives information on a different attitude to coping. The scores on the sub-scales allow an interpretation to be made of which attitude to coping an individual uses most.
The Coopersmith Self-Esteem Inventory | after three months
  The Coopersmith Self-Esteem Inventory was developed by Stanley Coopersmith(1986), and adapted to Turkish by Turan and Tufan(1987), who also carried out the validity and reliability study. It consists of 25 items, which contain statements about the person's outlook on life, family relations, social relations and endurance. Scores range from 0 to 100.